CLINICAL TRIAL: NCT01369251
Title: Simple Hygiene Versus Alcohol Based Usual Care for Umbilical Cord: a Randomized Clinical Trial
Brief Title: Simple Hygiene Versus Alcohol Based Usual Care for Umbilical Cord
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASST Fatebenefratelli Sacco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSaccoCordCare
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-04

CONDITIONS: Infection; Skin Diseases, Bacterial; Granuloma
MeSH Terms: conditions — Infections; Skin Diseases, Bacterial; Granuloma | interventions — Hygiene; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hygiene with water and soap (Experimental)
  Interventions: Behavioral: Hygiene
- Usual alcohol care (Active Comparator)
  Interventions: Procedure: Usual alcohol care

INTERVENTIONS:
Behavioral: Hygiene
  Arms: Hygiene with water and soap
Procedure: Usual alcohol care
  Arms: Usual alcohol care

SUMMARY:
The purpose of this study is to determinate whether in newborns just cleaning the umbilical stump when changing diapers (with water and soap if necessary)is effective in preventing local cord infections and not delaying cord separation as just as cord care alcohol, usually applied in our hospital and suggested to parents at dismission.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate for gestational age newborn

Exclusion Criteria:

* Not appropriate for gestational age newborn

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
omphalitis incidence

SECONDARY OUTCOMES:
umbilical granuloma incidence
time to cord separation

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Meroni, Study Director — ASST Fatebenefratelli Sacco; Maria Teresa Garavaglia, Study Chair — ASST Fatebenefratelli Sacco; Ludovica Tagliabue, MD, Principal Investigator — Università di Milano
Locations (1):
- Ospedale Luigi Sacco, Milan, Italy